CLINICAL TRIAL: NCT06682364
Title: Opioid Use and Criminal Justice: Intervening to Improve the Outcomes of Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abenaa Jones, Ph.D. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Abenaa Jones, Ph.D., Ann Atherton Hertzler Early Career Professor in Health and Human Development, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00023933; K01DA051715 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder
Keywords: women; criminal justice; substance use; opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case management using certified recovery specialists (Active Comparator): The arm incorporates several best practices in substance use treatment such as the use of Certified Peer Recovery Specialists (CRS) as needed social support, assisting women who do not have stable housing in finding housing, overdose response training, and reducing known barriers to women by assisting with transportation and childcare.
  Interventions: Behavioral: Trauma-informed case management for women who use drugs; Behavioral: CRS Only Intervention
- Case management using certified recovery specialists + Trauma Support Group (Experimental): Includes all the components in the comparative arm and a 12-session trauma support group led by CRS, which uses the evidence-based curriculum, Beyond Trauma, which was specifically designed for women who use drugs.
  Interventions: Behavioral: Trauma-informed case management for women who use drugs

INTERVENTIONS:
Behavioral: Trauma-informed case management for women who use drugs — This intervention assesses the adequacy in which components of the gender-specific and trauma-informed intervention function together using a sample of 50 community-recruited CJI women who use opioids illicitly.
Behavioral: CRS Only Intervention — This intervention assesses the adequacy in which components of the gender-specific case management by certified peer recovery specialists function together using a sample of 50 community-recruited CJI women who use opioids illicitly.
  Arms: Case management using certified recovery specialists

SUMMARY:
Opioid-related overdose deaths and incarceration rates have skyrocketed and have disproportionately affected women. Despite having a higher burden of substance use disorders and HIV/AIDS than criminal justice-involved (CJI) men, CJI women are less likely to have access to substance use and HIV treatment. The planned research aims to improve how women in the criminal justice system connect to and stay in drug treatment. This will be done by creating and putting into practice a well-researched program specifically designed for women, considering their experiences with trauma. The program incorporates several best practices in substance use treatment such as the use of Certified Peer Recovery Specialists (CRS) as needed social support, assisting women who do not have stable housing in finding housing, overdose response training, and reducing known barriers to women by assisting with transportation and childcare. In addition, half of the women will be randomly selected to participate in a 12-session trauma support group led by CRS which uses the evidence-based curriculum, Beyond Trauma, which was specifically designed for women who use drugs. The aforementioned components are rarely offered in tandem with substance use treatment, and as such, this research is assessing if having this comprehensive program is linked with better substance use and social outcomes. The overall goal is to reduce the problem of opioid addiction and overdoses among women who have recently been involved in the criminal justice system and to reduce the barriers to opioid addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18+ years of age
3. Pennsylvania resident and intends to remain in or near Harrisburg, Carlisle, York or Lancaster areas for the duration of the study
4. Use opioids illicitly
5. Interested in starting drug treatment that uses medication to stop opioid use OR are currently in a drug treatment program for opioid use that uses medication but feel that without additional support they won't be able to continue with the program
6. Not currently pregnant, planning to become pregnant, or breastfeeding during the study period
7. Released from a jail or prison within the past 12 months or have other criminal justice involvement (arrests, probation, or parole) within the past 12 months.

Exclusion Criteria:

1. Not female
2. Under 18 years of age
3. Not a Pennsylvania resident or no intention to remain in or near Harrisburg/Carlisle/York or Lancaster areas for the duration of the study
4. Do not use opioids illicitly
5. Not interested in MOUD to stop opioid use
6. No arrests, probation or parole, nor released from a jail or prison within the past 12 months
7. Pregnant, planning to become pregnant, or breastfeeding during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled and retained in the intervention | 6 months of follow-up for participants
  We will assess the feasibility of this pilot study by assessing the number of participants recruited and retained for the entire six-month duration of the intervention.

SECONDARY OUTCOMES:
Preliminary substance use outcomes | 6 months of follow-up for participants
  The investigators will assess participants' urine drug screen results at baseline, 3-month follow-up, and 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Abenaa Jones, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Recovery, Advocacy, Service, and Empowerment (RASE), Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be deposited into the National Addiction and HIV Data Archive Program
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The information will be available by the project end date or when the first paper based on the data is published, whichever is first.
Access Criteria: Investigators interested in using data and accessing the National Addiction & HIV Data Archive Program will have access to de-identified data from participants at all time points.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/index.html